CLINICAL TRIAL: NCT01611584
Title: A Proof of Principle Study of Aminolevulinic Acid (ALA) - Induced Fluorescence Detection in Resectable Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D1046
Record Dates: First submitted 2012-04-10; First posted 2012-06-05 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Lung Cancer in Normal and Malignant Tumors
Keywords: ALA; Florescence; Lung cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALA (Experimental): No arms for the trial. Participants will have proven or presumed lung cancer and will be assessed for participant by a research team member.
  Interventions: Drug: ALA-induced Fluorescence

INTERVENTIONS:
Drug: ALA-induced Fluorescence — ALA Dose- 20 mg/kg

SUMMARY:
The purpose of this trial is to measure ALA-induced fluorescence in both normal and malignant tissue.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria Patients (12 total patients with lung cancer) meeting eligibility criteria will be enrolled.
* Preoperative diagnosis of either presumed or documented non-small cell lung cancer.
* Tumor judged to be suitable for surgical resection based on preoperative evaluation of radiographic studies, pulmonary function tests, performance status and clinical judgment of surgeons at DHMC (Erkmen, Nugent)
* Age ≥ 18 years old.
* Population representative of our usual referral pattern including minority populations, women and those who are financially disadvantaged.
* Subjects capable of giving informed consent

Exclusion Criteria:

* Pregnant Women
* Women who are breast feeding
* History of cutaneous photosensitivity
* Porphyria, hypersensitivity to porphyrins, photodermatosis
* Exfoliative dermatitis
* History of liver disease within the last 12 months
* Inability to comply with photosensitivity precautions associated with the study
* Inability to give informed consent
* AST, ALT, ALP or bilirubin levels greater than 2.5 times the normal limit at any time during the past 2 months
* Plasma creatinine in excess of 180 umol/L
* Women who are breast feeding
* History of cutaneous photosensitivity
* Porphyria, hypersensitivity to porphyrins, photodermatosis
* Exfoliative dermatitis
* History of liver disease within the last 12 months
* Inability to comply with photosensitivity precautions associated with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
ALA-induced fluorescence- lung cancer | Participants will be followed for duration of the hospital stay, and up to 3 weeks after
  Determine the relationship between ALA induced protoporphyrin IX (PplX) flourescence and histology in both normal and malignant tumors.

SECONDARY OUTCOMES:
Determine Feasibility of fluorescence | Participants will be followed for the duration of their hospital study and up to 3 weeks after
  Determine feasibility of integrating fluorescence detection into surgical pratice of resection for lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Cherie P Erkmen, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States